CLINICAL TRIAL: NCT02724436
Title: Radioembolization With Yittrium-90 for Intermediate and Advanced Hepatocellular Carcinoma: A Randomized Controlled Trial
Brief Title: Radioembolization With Yittrium-90 for Intermediate and Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012ZX10002016003002
Record Dates: First submitted 2016-03-28; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma; Radioembolization
Keywords: Yittrium-90; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Yttrium-90

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TACE (Experimental): transcatheter arterial chemoembolization
  Interventions: Procedure: TACE
- TACE+radioembolization (Experimental): TACE plus radioembolization with Y-90: 100
  Interventions: Procedure: TACE; Procedure: radioembolization with Y-90

INTERVENTIONS:
Procedure: TACE
Procedure: radioembolization with Y-90 — radioembolization with Y-90
  Arms: TACE+radioembolization

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most-common cancer worldwide and the second most-common cause of cancer mortality. Liver resection is the first-line curative treatment for huge HCC. The 5-year overall survival (OS) rates after hepatic resection were range from 25% to 45%. Transarterial chemoembolization (TACE) is the major treatment option for the unresectable primary or secondary liver malignancies. Yittrium-90 (Y-90) is a pure beta-emitter, without any toxic effect or immune rejection. There are ample data that support the use of Y-90 microspheres for primary and metastatic liver tumors. The aim of our study was to compare the clinical outcome of radioembolization with Y-90 and TACE and provide a new strategy for the treatment of intermediate and advanced hepatocellular carcinoma with portal vein thrombus by conduting a randomized trial.

ELIGIBILITY:
Inclusion Criteria:

1. Child-Pugh class A or B liver function;
2. Preoperative ECOG criteria score of 0-2;
3. Patients preoperatively diagnosed of hepatocellular carcinoma according to chest computed tomography (CT) and/or magnetic resonance imaging (MRI);
4. Tumor number ≤5 and the sum of largests tumor diameter ≤15 cm;
5. The expected survival time >6 months.

Exclusion Criteria:

1. Other anticancer treatment before treatment
2. Patients with apparent major organs (i.e. cardiac, pulmonary, cerebral and renal) dysfunction, which may affect the treatment of liver cancer
3. Patients with other diseases that may affect the treatment of this treatment
4. History of other malignant tumors
5. Patients who are participating in other clinical trials
6. Pregnant, lactating women

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years
Time to progress | 3 years
Toxic and side effects caused by TACE or radioembolization with Y-90 | 3 years
Postoperative complication | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China